CLINICAL TRIAL: NCT03864029
Title: An Observational Study Research to Collect the Effectiveness and Safety Data of KUVAN® Retrospectively in Chinese Subjects With Hyperphenylalaninemia (HPA) Caused by Tetrahydrobiopterin (BH4) Deficiency
Brief Title: Retrospective Observational Safety Effectiveness With Kuvan in hpA
Acronym: ROSEKA
Status: Completed | Type: Observational
Sponsor: BioMarin Pharmaceutical (Industry)
Collaborators: Quintiles, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: BMN 162-504
Record Dates: First submitted 2019-02-22; First posted 2019-03-06 (Actual); Last update posted 2019-03-07 (Actual); Status verified 2019-03

CONDITIONS: Tetrahydrobiopterin Deficiency
MeSH Terms: conditions — Phenylketonurias | interventions — sapropterin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

INTERVENTIONS:
Drug: KUVAN — retrospective data on the effectiveness of past treatment with KUVAN®. It includes blood Phe level, physical development status, intelligence development status, etc., during treatment with KUVAN
  Other Names: Diagnostic Tests

SUMMARY:
A retrospective study to collect the effectiveness and safety data of the past treatment with KUVAN in Chinese patients with HPA caused by BH4 deficiency. The data was collected from relevant past medical history and past clinical and safety assessments.

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to provide informed consent (unless exemption of obtaining consent is obtained as per local regulation). Assent (if required defined by local regulation and requirement) should also be obtained from the subject and the legal authorized representative.
* Diagnosed with BH4 deficiency per local practice.
* KUVAN® was taken at least 1 dose to treat HPA caused by BH4 deficiency during the period of observation.
* Baseline Phe concentration ≥ 450 µmol/L

Exclusion Criteria:

* Subject diagnosed to have Phenylketonuria (PKU)
* Has any condition that, in the view of the Investigator, the medical record of the subject in the duration of observation is not reliable, or not accessible.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Chinese subjects with HPA caused by BH4 deficiency
Sampling Method: Non-Probability Sample
Enrollment: 26 (Actual)
Dates: Start 2017-10-10 (Actual); Primary Completion 2018-03-09 (Actual); Study Completion 2018-07-25 (Actual)

PRIMARY OUTCOMES:
Diagnosis on BH4 deficiency based on medical history - laboratory testing results indicating sub-type (% in each sub-type) • Incidents and severity of AE reported (% of incident / % of each severity) | 2010-2015
Retrospective KUVAN treatment history - dose (mg/kg/day), | 2010-2015
Retrospective KUVAN treatment history - length of exposure (days) | 2010-2015
Retrospective Baseline Phe concentration ≥ 450 μmol/L - laboratory testing results (μmol/L) | 2010-2015
Number of participants with AE reported (% of patient with AE reported) | 2010-2015
Incidents and severity of AE reported (% of incident / % of each severity) | 2010-2015
Retrospective blood Phe level as indicated in laboratory testing results (μmol/L) | 2010-2015
Retrospective body height as indicated in medical note (cm) | 2010-2015
Retrospective body weight as indicated in medical note (kg) | 2010-2015
Retrospective occipital / frontal circumferences as indicated in medical note (cm) | 2010-2015
Retrospective intelligence development status via China local standard development assessment method (score) | 2010-2015

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, MD, Study Director — Medical Director
Locations (1):
- West China Hospital of Sichuan University, Chengdu, Sichuan, China